CLINICAL TRIAL: NCT04162717
Title: The Effect of Telephone Symptom Triage Protocols on Symptom Management, Quality of Life and Self-Care Maintenance in Patients With Cancer Who Applied Systemic Treatment: A Randomized Controlled Trial
Brief Title: The Effect of Telephone Symptom Triage Protocols in Patients With Cancer Therapy (TeleTRIAGE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Arife ALTIN ÇETİN, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0010
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Cancer; Self Efficacy
Keywords: Patients with cancer; Symptom triage; Self care; Symptom management; Quality of life
MeSH Terms: conditions — Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Telephone Symptom Triage Protocols (Experimental): Intervention group received symptom triage application with telephone, which consisted of guiding in line with symptom triage protocols. The patients who were included in the intervention were followed up by telephone on the 3rd, 7th and 10th day of after chemotherapy total of nine times during three chemotherapy cycles.
  Symptom management, quality of life and self-maintenance were assessed by scales at the first interview and 3 months later.
  Interventions: Behavioral: The Effect of Telephone Symptom Triage Protocols on Symptom Management, Quality of Life and Self-Care Maintenance in Patients with Cancer Who Applied Systemic Treatment
- Control group (No Intervention): The control group received standard nursing care applied at the hospital

INTERVENTIONS:
Behavioral: The Effect of Telephone Symptom Triage Protocols on Symptom Management, Quality of Life and Self-Care Maintenance in Patients with Cancer Who Applied Systemic Treatment — Symptom management, quality of life and self-maintenance were assessed by scales at the first interview and 3 months later.
  Intervention group received symptom triage application with telephone, which consisted of guiding in line with symptom triage protocols. The patients who were included in the intervention were followed up by telephone on the 3rd, 7th and 10th day of after chemotherapy total of nine times during three chemotherapy cycles.
  Arms: The Effect of Telephone Symptom Triage Protocols

SUMMARY:
The purpose of this study was to evaluate the effect of telephone symptom triage protocols on symptom management, quality of life and self-maintenance in patients with cancer who applied systemic treatment. The study is a randomized controlled experimental study. Pan-Canadian Oncology Symptom Triage and Remote Support (COSTaRS) guides were translated into Turkish and expert opinions were obtained. The sample of the study included 70 cancer (35 interventions and 35 controls) patients who were treated with chemotherapy were randomized into the computer program.

According to the interference protocol of the study: Preliminary interviews were conducted with the newly diagnosed patients in the control and intervention groups. Preliminary tests (Personal Information Form, Chemotherapy Symptom Assessment Scale, Functional Assessment of Cancer Therapy Form-General - FACT-G (Version 4) Quality of Life Scale and Self-Care Power Scale) were performed after obtaining consent. After the pre-tests, the patients who were included in the intervention group were given the symptom triage protocol usage guide created according to the symptom triage protocol. The patients were informed by the researcher about the content and use of the guideline. The patients included in the intervention group were searched by the researcher on the 3rd, 7th and 10th days after each chemotherapy for 3 cycles of chemotherapy. During the three-month follow-ups, patients were able to call the investigator 7/24 to request symptom triage. In accordance with the Remote Symptom Management Guidelines for Adults Treated with Cancer, patient triage was performed for symptom management and patients were referred to the appropriate sources according to the severity of the symptom. The patients in the control group did not undergo any intervention other than routine hospital follow-up. Patients who were included in the control and intervention groups were subjected to final tests at the hospital after 3 months.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of telephone symptom triage protocols on symptom management, quality of life and self-maintenance in patients with cancer who applied systemic treatment. The study is a randomized controlled experimental study.

Before starting the research, permissions were taken. Pan-Canadian Oncology Symptom Triage and Remote Support (COSTaRS) guides were translated into Turkish and expert opinions were obtained.

The sample of the study included cancer patients who were treated with chemotherapy in the Akdeniz University Hospital Day Chemotherapy Unit. The study included 80% power, 95% reliability and 0.05 error margins, and 70 patients (35 interventions and 35 controls) were randomized into the computer program.

According to the interference protocol of the study:

* Four patients who received systemic chemotherapy were tested with pilot study.
* Patients were included in the study according to the inclusion criteria and randomization list.
* Preliminary interviews were conducted with the newly diagnosed patients in the control and intervention groups. Preliminary tests were performed after obtaining consent. For this purpose, Personal Information Form, Chemotherapy Symptom Assessment Scale, Functional Assessment of Cancer Therapy Form-General - FACT-G (Version 4) Quality of Life Scale and Self-Care Power Scale were applied.
* After the pre-tests, the patients who were included in the intervention group were given the symptom triage protocol usage guide created according to the symptom triage protocol. The patients were informed by the researcher about the content and use of the guideline. Information about the contents of the guide was made between 10:00-14:00 hours during working hours during the week and it took an average of 15-20 minutes.
* The patients included in the intervention group were searched by the researcher on the 3rd, 7th and 10th days after each chemotherapy for 3 cycles of chemotherapy.
* During the three-month follow-ups, patients were able to call the investigator 7/24 to request symptom triage.
* In accordance with the Remote Symptom Management Guidelines for Adults Treated with Cancer, patient triage was performed for symptom management and patients were referred to the appropriate sources according to the severity of the symptom.
* In case of urgent necessity, patients were referred from the second consultant who were from Medical Oncology Department.
* The frequency of calls for the symptom triage protocol application of the intervention group was monitored and the information was recorded in the intervention group telephone interview form.
* The patients in the control group did not undergo any intervention other than routine hospital follow-up.
* Patients who were included in the control and intervention groups were subjected to final tests at the hospital after 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Able to come to Medical Oncology Polyclinic and Chemotherapy Unit for outpatient treatment
2. First-time diagnosed cancer
3. Know her/his diagnossis and/or able to express verbal
4. Having undergone a cure chemotherapy treatment
5. Chemotherapy was applied every 21-28 days
6. Between 18-65 years (not to interfere with physical, psychological and functional problems that may develop due to old age)
7. Able to understand and write Turkish
8. Able to use mobil telephone
9. No disability to answer questions physically, cognitively or spiritually
10. Non-bed dependent
11. Willing to participate

Exclusion Criteria:

1. Having diagnosed with psychiatric disease
2. Having memory or cognitive disorder
3. Patients receiving chemotherapy every seven or 14 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Chemotherapy Symptom Assessment Scale (C-SAS) | 12 week
  The scale was developed by Brown et al. (2001) in the UK and aims to measure 24 chemotherapy symptoms in cancer patients receiving chemotherapy. C-SAS consists of three parts.The highest and lowest scores are not calculated for the total score in the scale. Since each symptom is evaluated separately, the median values are calculated instead of the arithmetic mean. In this study, Turkish version of the scale was used.
Functional Assessment of Cancer Therapy Forum-General - FACT-G (Version 4) | 12 week
  The scale was developed by "Center on Outcomes, Research, and Education Northwestern Healthcare" in USA and it is used to evaluate the quality of life of malignant patients.The FACT-G assesses four dimensions of quality of life: physical status, social and family status, emotional status and activity status.The FACT-G contains 27 items and each item score ranges from 0 to 5.The total score is between 0-108. High score indicates that the individual perceives life quality is to be high. In this study, Turkish version of the scale was used.
The self-care agency scale | 12 week
  The scale was developed by Kearney ve Fleicher (1979) to measure people's ability to look after themselves or their power. The scale contains 35 items and each item score ranges from 0 to 5. The highest and lowest possible score is between 35-140. The scores according to the Self-Care Agency scale is considered 24-64 points are as poor, 65-100 points as moderate, 101-112 points as good and 113-138 points as very good self-care power level. The higher scores indicates better self-care ability of the individual. In this study, Turkish version of the scale was used.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran BEKTAŞ, Professor, Study Chair — Akdeniz University Faculty of Nursing
Locations (1):
- Arife Altin Cetin, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cetin AA, Bektas H, Coskun HS. The effect of telephone triage on symptom management in patients with cancer undergoing systemic chemotherapy: A randomized controlled trial. Eur J Oncol Nurs. 2022 Dec;61:102221. doi: 10.1016/j.ejon.2022.102221. Epub 2022 Oct 13. PMID 36332454